CLINICAL TRIAL: NCT01954979
Title: A Phase I Study of Abatacept in the Treatment of Patients With Steroid Refractory Chronic Graft Versus Host Disease (cGVHD)
Brief Title: Abatacept to Treat Steroid Refractory Chronic Graft Versus Host Disease (cGVHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jacalyn Rosenblatt, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-358
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Graft versus Host Disease; ABATACEPT
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abatacept (Experimental): Abatacept will be administered for a total of 6 doses. Doses 1-3 will be administered at two week intervals (+/-2 days). One month following Dose 3, abatacept will be administered, and given at four-week intervals (+/-2 days) for three doses (Doses 4-6.) Patients will be followed for toxicity for 28 days following last dose of Abatacept. Patients will then be seen monthly for six months.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — The study will follow a standard 3+3 design with two escalating doses of abatacept to determine the maximum tolerated dose (MTD): 3 mg/kg (dose level 1) and 10 mg/kg (dose level 2). Dose-limiting toxicities (DLTs) are defined as any Grade 3 or 4 toxicities judged to be probably or definitely related to abatacept.

SUMMARY:
The participant is invited to take part in this study because they have chronic Graft versus Host Disease (cGVHD) that is not responding to standard treatment with steroids. This research study is a way of gaining new knowledge about the treatment of patients with cGVHD. This research study is evaluating a drug called abatacept.

Abatacept is a drug that alters and suppresses the immune system. Abatacept is approved by the Food and Drug Administration (FDA) for the treatment of moderate to severe active rheumatoid arthritis in adults and of severe juvenile idiopathic arthritis (JIA) in patients who have failed prior therapy with disease-modifying anti-rheumatic drugs (DMARDs). These are autoimmune conditions, ie caused by an overactive immune system that attacks normal tissues and organs. It is currently being tested in a variety of other autoimmune conditions. In this case it is considered experimental.

cGVHD is caused by the donor cells attacking various organs of the recipient. The investigators try to minimize this immune attack by using corticosteroids such as prednisone. In severe cases prednisone is not sufficient and other immunosuppressive medications are used in addition in order to more efficiently control cGVHD and to limit the dose and consequently the multiple side-effects of corticosteroids. This study is being done to determine if the use of abatacept is safe in patients with cGVHD and if it can facilitate a better control of cGVHD.

During this study the participants will be evaluated for side effects from the treatment with abatacept, and for response of the cGVHD to the treatment. There will be two groups of participants in the study. The first group will be treated at a relatively low dose of abatacept. If this is found to be safe then the second group will be treated at a higher dose. Three to four tablespoons of blood will be drawn at every 2 week visit in order to determine your blood counts, kidney and liver function. Some of the blood will be used in a research lab in order to study measures of your immune system and how they might be affected by the treatment.

DETAILED DESCRIPTION:
Before the research starts (screening): After signing the consent form, the participant will be asked to undergo some screening tests or procedures to find out if they can be in the research study. Many of these tests and procedures are likely to be part of regular cGVHD care and may be done even if it turns out that the participant does not take part in the research study. If the participant has had some of these tests or procedures recently, they may or may not have to be repeated.

* Complete Medical History and Physical Examination
* Blood Collection: 3-4 tablespoons of blood will be drawn to measure the participants complete blood counts, kidney, liver and thyroid function
* Disease Assessment: Depending on what organs are affected by their cGVHD the participant may undergo blood tests or a skin exam or an eye exam or a dental exam.
* Electrocardiogram (EKG): a noninvasive test that measures the electrical activity of the participant's heart
* A tuberculin skin test and a quantiferon blood test to rule out tuberculosis
* Pregnancy testing if applicable
* HIV and Hepatitis blood test: 2-3 teaspoons of blood will be collected to perform an HIV test. The participant will be asked to sign a separate consent form for this test. The participant's doctor will discuss the results of this test with the participant and the results will become a part of their permanent medical record. The participant may seek private HIV testing prior to consenting, and based on the results may choose whether or not to participate in this study or have the HIV test become part of their medical records.

If these tests show that the participant is eligible to participate in the research study, the participant will begin the study treatment. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.

Additional research procedures to be performed at the time of screening:

- Research blood testing: to study measures of the participant's immune system

After the screening procedures confirm that the participant is eligible to participate in the research study:

* Since the investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have abatacept, not everyone who participates in this research study will receive the same dose of the study drug. The dose the participant gets will depend on the number of participants who have been enrolled in the study before the participant and how well they have tolerated their doses.
* The total duration of treatment on this study is approximately 113 days or 6 treatments. Doses 1-3 will be administered every two weeks. One month following Dose 3, abatacept will be administered every four weeks for the remaining three doses (Doses 4-6.) The treatment will be given intravenously on these days. One month following your last dose of treatment, the participant will be seen in clinic. The participant will be seen in the clinic weekly through dose 4, then every 2 weeks for follow up even if the participant doesn't have treatment.
* The first group of participants will be treated with a lower dose of abatacept. If this dose is determined to be safe then the second group will be treated at a higher dose.

During treatment the participant will be seen in the clinic every two weeks. At every visit the following will be performed:

* Complete Medical History and Physical Examination
* Blood Collection: 3-4 tablespoons of blood will be drawn to measure their complete blood counts, kidney, liver and thyroid function
* Research blood testing: to study measures of the participant's immune system
* On the days of treatment the participant will undergo an assessment of cGVHD depending on what organs are affected

After the final dose of the study drug:

After the participant has completed taking the drug on the study, the following procedures and tests will take place:

* Safety assessment 28 days after the last dose of the study drug.
* Complete Medical History and Physical Examination
* Blood Collection: 3-4 tablespoons of blood will be drawn to measure the participant's complete blood counts, kidney, liver and thyroid function
* Disease Assessment: by physical exam and blood tests if the participant has leukemia or multiple myeloma, or physical exam and PET/CT or CT scan if the participant has lymphoma. These will be done at the safety assessment visit and at the 3 and 6 month follow up visits.
* Electrocardiogram
* Research blood testing: to study measures of your immune system
* Once the participant has completed treatment on study they will be followed monthly for 6 months

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Participants must be recipients of an allogeneic bone marrow or stem cell transplantation with myeloablative or reduced intensity conditioning regimens.
* Participants must be at least 100 days after the transplantation or a donor lymphocyte infusion.
* Participants must have cGVHD (as defined by the National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease)
* Participants may have either extensive or limited cGVHD requiring systemic treatment
* Participants must have steroid refractory cGVHD, defined as having persistent signs and symptoms of chronic GVHD despite the use of prednisone at ≥ 0. 5 mg/kg/day (or equivalent) for at least 4 weeks in the preceding 12 months. Patients may remain on steroids while enrolled in the study.
* No addition or subtraction of other immunosuppressive medications for at least 4 weeks prior to starting treatment.
* On stable immunosuppressive regimen for 2 weeks prior to enrollment. Adjustment of immunosuppressive medications to maintain a therapeutic level is permitted.
* Age ≥ 18 years at the time of signing the informed consent form.

Reproductive Status: Definition of Women of Child-Bearing Potential (WOCBP). WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal (see definition below).

Post-menopause is defined as:

* Women who have had amenorrhea for ≥ 12 consecutive months (without another cause) and who have a documented serum follicle-stimulating hormone (FSH) level > 35 mIU/mL.
* Women who have irregular menstrual periods and a documented serum FSH level > 35 mIU/mL.
* Women who are taking hormone replacement therapy (HRT).

The following women are WOCBP:

* Women using the following methods to prevent pregnancy: Oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as intrauterine devices or barrier methods (diaphragm, condoms, spermicides).
* Women who are practicing abstinence.
* Women who have a partner who is sterile (eg, due to vasectomy). WOCBP must be using an acceptable method of contraception to avoid pregnancy throughout the study and for up to 10 weeks after the last dose of study drug in such a manner that the risk of pregnancy is minimized.
* WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 0 to 48 hours before the first dose of study drug.
* Women must not be breast-feeding.
* Sexually active fertile men must use effective birth control if their partners are WOCBP.
* Life expectancy of greater than > 3 months.
* ECOG performance status ≤ 2 (see Appendix A).
* Laboratory test results within these ranges:
* Absolute neutrophil count ≥ 1500/mm³
* Serum creatinine ≤ 2.0 mg/dL
* Renal function assessed by calculated creatinine clearance ≥ 60ml/min by Cockcroft-Gault formula (see Appendix B: Cockcroft-Gault estimation of CrCl).
* Total bilirubin ≤ 1.5 x ULN (unless hepatic dysfunction is caused by cGVHD)AST (SGOT) and ALT (SGPT) ≤ 3 x ULN (unless hepatic dysfunction is caused by cGVHD).
* Patients much have a negative PPD skin test and a negative Quantiferon assay.
* Must possess the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Any serious medical condition (including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia), laboratory abnormality, or psychiatric illness/ social situation that would prevent the subject from signing the informed consent form or limit compliance with study requirements.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of starting treatment with abatacept.
* Use of biologic antibody therapy for cGVHD with rituximab, alemtuzumab, or ATG within 6 months of starting treatment with abatacept.
* Use of TNF alpha inhibitors within four weeks prior to study entry.
* Ongoing prednisone requirement >1 mg/kg/day (or equivalent)
* New immunosuppressive medication or ECP within 28 days of starting treatment with abatacept.
* Donor lymphocyte infusion within 100 days prior to enrollment.
* Active malignant disease relapse or other active malignancy with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Known seropositive for or positive viral load for HIV or positive viral loads for infectious hepatitis, type B (HBV) or C (HCV).
* Uncontrolled intercurrent active infection. Controlled infection on long term suppressive or maintenance therapy is permissible.
* Use of live vaccines within four weeks of starting abatacept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Determination of the Maximum Tolerated Dose (among two dose levels) and toxicity profile of a 141 day/6 dose course of abatacept in patients with steroid refractory cGVHD. | 2 Years
  Determination of the Maximum Tolerated Dose (among two dose levels) and toxicity profile of a 141 day/6 dose course of abatacept in patients with steroid refractory cGVHD.

SECONDARY OUTCOMES:
Determination of the efficacy (in terms of cGVHD symptoms, score and steroid dose) of a 141 day/6 dose course of abatacept in patients with steroid refractory cGVHD | 2 Years
  Determination of the efficacy (in terms of cGVHD symptoms, score and steroid dose) of a 141 day/6 dose course of abatacept in patients with steroid refractory cGVHD
Examination of the immunologic effects associated with the administration of abatacept in patients with steroid refractory cGVHD. | 2 Years
  Examination of the immunologic effects associated with the administration of abatacept in patients with steroid refractory cGVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Rosenblatt, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Koshy AG, Kim HT, Liegel J, Arnason J, Ho VT, Antin JH, Joyce R, Cutler C, Gooptu M, Nikiforow S, Logan EK, Elavalakanar P, Narcis M, Stroopinsky D, Avigan ZM, Boussi L, Stephenson S, El Banna H, Bindal P, Cheloni G, Avigan DE, Soiffer RJ, Rosenblatt J. Phase 2 clinical trial evaluating abatacept in patients with steroid-refractory chronic graft-versus-host disease. Blood. 2023 Jun 15;141(24):2932-2943. doi: 10.1182/blood.2022019107. PMID 36862975
- [Derived] Nahas MR, Soiffer RJ, Kim HT, Alyea EP 3rd, Arnason J, Joyce R, Antin JH, Ho VT, Stroopinsky D, Li S, Levine JD, McMasters M, Jain S, Hamdan A, Tzachanis D, Bryant MP, Logan EK, Bazemore J, Stewart J, Joyce A, Stephenson S, Washington A, Cole L, Pyzer A, Leaf RK, Avigan DE, Rosenblatt J. Phase 1 clinical trial evaluating abatacept in patients with steroid-refractory chronic graft-versus-host disease. Blood. 2018 Jun 21;131(25):2836-2845. doi: 10.1182/blood-2017-05-780239. Epub 2018 Mar 16. PMID 29549175